CLINICAL TRIAL: NCT03642587
Title: Canadian Sudden Cardiac Arrest Network
Acronym: C-SCAN
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Collaborators: University of Toronto (Other); Sunnybrook Health Sciences Centre (Other); Ottawa Hospital Research Institute (Other); University of British Columbia (Other); Providence Health & Services (Other); McMaster University (Other); Queen's University, Kingston, Ontario (Other); Institute for Clinical Evaluative Sciences (Other); Alberta Health services (Other); University of Saskatchewan (Other); Dalhousie University (Other); University of Prince Edward Island (Other); Memorial University of Newfoundland (Other)
Responsible Party: Sponsor
Other Study IDs: CSCAN version 2
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Sudden Cardiac Death; Sudden Cardiac Arrest
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Population: People between the ages of 2 and 85 years old with out of hospital cardiac arrest of no obvious cause who are attended to by paramedics who survive or die
  Interventions: Other: There is no intervention in this study.

INTERVENTIONS:
Other: There is no intervention in this study. — There is no intervention in this study.

SUMMARY:
The overall aim of the project is to develop a national registry to accurately measure the burden of Sudden Cardiac Arrest (SCA) among the general Canadian population. This project will create a common platform to link existing sources of information (EMS, Coroner and Administrative Databases) in order to fully understand the causes and outcomes of SCA. This comprehensive, unique registry will inform the progress and effectiveness of all CANet SCA programs aimed at reducing SCA. Understanding the antecedents, causes and outcomes of SCA will allow for new initiatives/investigations to reduce SCA, by using targeted interventions both effectively and efficiently.

DETAILED DESCRIPTION:
SCA is defined as an abrupt collapse with documented loss of vital signs,in a seemingly healthy individual and attributable to a cardiac cause. Estimates of SCA incidence vary widely from 53 to 153 per 100,000 persons/year. Most published studies use public reporting, death certificates or autopsy based registries to identify and classify SCA cases, but limited sources often result in missed cases. Prospective registries monitoring SCAs over time in large populations provide the most accurate estimation of incidence rates.

An ongoing challenge in developing effective strategies to decrease SCA are the varying definitions used to define SCA. Many published studies identify SCA as OHCA of "no obvious cause" (assumed to be a cardiac arrest due to an underlying primary cardiac cause); however, the two are not synonymous. Verifying that a particular OHCA is due to cardiac disease requires careful establishment, using data from multiple sources and case-by-case adjudication, which is difficult and not routinely performed. Accurate identification of true SCAs is crucial if we plan to implement interventions aimed to prevent them.

The Canadian Resuscitation Outcomes Consortium (CanROC) investigators are proposing to leverage experience gained from developing a sophisticated registry of all emergency medical service (EMS)-attended OHCA patients in Ontario and British Columbia (Resuscitation Outcomes Consortium - ROC 2005-2015). This registry has since been spread across Canada to include nine other provinces covering >15 million people in urban and rural communities. The proposed C-SCAN Registry will leverage and expand upon the CanROC infrastructure by augmenting its dataset to include detailed information both preceding and following the SCA event. Using this information to identify high-risk patients, we aim to implement targeted initiatives to decrease the incidence of SCA in Canada.

Objectives:

1. To accurately identify and classify all possible SCA cases within the study area using new and existing data sources.
2. To accurately measure the incidence and causes of SCA by age and sex.
3. To measure the triggers and warning signs of SCA cases in relation to age, sex and etiology for the purposes of prediction and prevention.
4. To confirm if the preliminary/pilot observations seen in southern Ontario are mirrored in other Canadian communities, both urban and rural, and in communities that are culturally and ethnically different from those in urban Toronto.

ELIGIBILITY:
Inclusion Criteria:

* All out of hospital cardiac arrest cases of "no obvious cause"
* Age between 2 and 85 years
* Attended to by paramedics, and survived or died.

Exclusion Criteria:

* Patients under the age of 2 years old or older than the age of 85 years old
* Do not resuscitate orders
* Cardiac arrests with obvious causes such as trauma, anaphylaxis, sudden upper airway occlusion, asthma, confirmed drug overdoses, homicides and suicides.

Ages: 2 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People between the ages of 2 and 85 years old with out-of-hospital cardiac arrest of no obvious cause who are attended to by paramedics who survive or die.
Sampling Method: Non-Probability Sample
Enrollment: 82054 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Incidence of SCA | 2 years
  Incidence of sudden cardiac arrest across Canada, by province, age and sex

CONTACTS AND LOCATIONS:
Overall Officials: Steve S Lin, MD, MSc, Principal Investigator — Unity Health Toronto
Locations (6):
- Canada (6):
  - Alberta Health Services, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Emergency Health Services, Halifax, Nova Scotia
  - Ottawa Health Research Institute, Ottawa, Ontario
  - Urgences-Sante, Montreal, Quebec
  - Saskatchewan Health Authority, Saskatoon, Saskatchewan